CLINICAL TRIAL: NCT03920800
Title: Preventing Invasive Cervical Cancer: The Importance of Expectant Management in Young Women With High-grade Pre-cancerous Lesions
Status: Completed | Type: Observational
Sponsor: Catherine Vanpachterbeke (Other)
Responsible Party: Sponsor-Investigator, Catherine Vanpachterbeke, Head of clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-Salem Wehbe
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: High-Grade Squamous Intraepithelial Lesions
MeSH Terms: conditions — Squamous Intraepithelial Lesions | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — * Pap smear
  * Cervical biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Conservative management - progression: Young women with high grade pre-cancerous lesions, followed within the CHU Brugmann Hospital according to a conservative attitude, with progressive lesions or lesions remaining present after 2 years of follow-up.
  Interventions: Other: Data extraction from medical files; Biological: Immunohistochemistry
- Conisation: Young women with high grade pre-cancerous lesions, followed within the CHU Brugmann Hospital by means of conisations.
  Interventions: Other: Data extraction from medical files; Biological: Immunohistochemistry
- Conservative management - spontaneous regression: Young women with high grade pre-cancerous lesions, followed within the CHU Brugmann Hospital according to a conservative attitude, who showed a spontaneous regression of the lesions during the 2 years follow-up.
  Interventions: Other: Data extraction from medical files; Biological: Immunohistochemistry

INTERVENTIONS:
Other: Data extraction from medical files — Data extraction from medical files
Biological: Immunohistochemistry — Immunohistochemistry with Ki67 and p16 antibodies on residual samples, if this had not been foreseen in the standard of care management of the patient.

SUMMARY:
Lesions classified as "High Grade Squamous Intra-epithelial Lesions" (HSIL) are pre-cervical lesions of the cervix, induced by infection with the Human Papilloma Virus (HPV). The detection and proper management of these lesions greatly reduces the incidence of invasive cervical cancer.

Pap smear remains the most effective tool for early detection of low and high-grade cervical lesions. In Belgium, screening for cervical cancer is recommended every 3 years for women between 25 and 65 years old.

HPV is a virus who possesses certain oncogenic genes who have the ability to inactivate tumor suppressor genes in the host cell. This promotes a tumorigenesis process within the tissues affected by the virus. The majority of human papillomavirus infections are transient and spontaneously cleared by host defense mechanisms, especially in the first two years after exposure. However, 10-20% of infections persist latently and may eventually lead to progression to invasive cervical cancer.

Even high-grade lesions kan naturally be cleared, even more so if the patient is young and immuno-competent. Therefore, the management of HSIL lesions in young women has been modified and consists of adopting mainly a conservative attitude, with controls every 6 months for 2 years. This management makes it possible to avoid unnecessary conizations of the cervix which, in young nulliparous patients, are not devoid of heavy obstetric consequences during subsequent pregnancies (premature birth, perinatal mortality). Cervical conization will only be considered for lesions that progress during follow-up or that persist beyond 2 years. However, this type of follow-up requires that patients be compliant.

Our study has two main objectives:

* to determine the compliance of CHU Brugmann Hospital patients who have been proposed a conservative strategy for the management of HSIL lesions.
* to identify the predictive factors for the persistence and / or progression of high-grade pre-cancerous dysplastic lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed within the CHU Brugmann Hospital (no private practices).
* HSIL lesions confirmed by anatomopathologic analysis on cervical biopsies or cone specimen without evidence of invasive lesions

Exclusion Criteria:

* Invasive lesions

Ages: 18 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: Young women followed within the CHU Brugmann Hospital for HSIL lesions.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Patient observance | Every six months over a period of 24 months
  Numeric value: 1 (optimal), 2 (acceptable), 3 (absent).
  Groups having benefited from a conservative attitude: Optimal compliance: 4 consultations in 24 months and / or indication of conization. Acceptable compliance: 2 to 3 consultations in 24 months. Observance absent: 0 to 1 consultation in 24 months. Groups having benefited from conization:
  Optimal compliance: 2 consultations after conisation. Acceptable compliance: 1 after consultation. Observance absent: 0 consultation after conisation.
Cytologic results of the cervico-uterine smear. | Every six months over a period of 24 months
  Cytologic results of the cervico-uterine smear. Diagnose established by the anatomo-pathologist.
Histologic results of the cervical biopsies | Every six months over a period of 24 months
  Histologic results of the cervical biopsies.Diagnose established by the anatomo-pathologist.
Extent of dysplastic lesions | Every six months over a period of 24 months
  Defined as the number of quadrants reached by the lesion.
Endocervix damage | Every six months over a period of 24 months
  Is the endocervix affected by the HSIL lesion (yes or no) ?
Immuno-histologic results Ki67 | Every six months over a period of 24 months
  Percentage of Ki67 antibody reactivity on the cervix biopsies
Immuno-histologic results p16 | Every six months over a period of 24 months
  Percentage of p16 antibody reactivity on the cervix biopsies

SECONDARY OUTCOMES:
Gestity | Every six months over a period of 24 months
  Total number of pregnancies
Parity | Every six months over a period of 24 months
  Total number of children born
Age at first patient visit | 1 day
  Age at first patient visit
HIV status | Every six months over a period of 24 months
  HIV positive or negative
Smoking status | Every six months over a period of 24 months
  Smoking or non smoking
Response time to the convocation for colposcopy | Up to 24 months
  Time between the patient's appointment and the receipt of the convocation for colposcopy
HPV status | Every six months over a period of 24 months
  Positive or negative for HPV virus
Quality of colposcopic examinations | Every six months over a period of 24 months
  Defined as satisfactory or unsatisfactory (junction area completely seen or not seen).

CONTACTS AND LOCATIONS:
Overall Officials: Georges Salem Wehbe, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No